CLINICAL TRIAL: NCT06570057
Title: Engagement of coMmunity Through Participatory Learning and Action for cOntrol and preVEntion of Type II Diabetes and Its Risk Factors [EMPOWER-D]: Feasibility Trial in Urban Pakistan
Brief Title: Feasibility Trial in Urban Pakistan for Community Engagement in Preventing Type II Diabetes and Risk Factors
Acronym: EMPOWER-D
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baqai Institute of Diabetology and Endocrinology (Other)
Collaborators: University of York (Other); Khyber Medical University Peshawar (Other); HealthNet TPO (Other); National Institute for Health Research, United Kingdom (Other Government); Aga Khan University Hospital, Pakistan (Other)
Responsible Party: Principal Investigator, Abdul Basit, Professor, Baqai Institute of Diabetology and Endocrinology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EMPOWERD-FT-UPK-2022
Record Dates: First submitted 2024-08-16; First posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Type II Diabetes Mellitus
Keywords: Community-Based Participatory Research; Participatory Learning and Action Research; Type II Diabetes Mellitus; Intermediate hyperglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: Two-arm parallel study design would be used. Six clusters will be randomly selected from purely urban blocks of Karachi. The study sites will be selected in a manner that the risk of possible contamination between control and intervention groups is avoided. The intervention clusters will receive the 18-months long PLA intervention along with study assessments, while the control clusters will only go through assessments i.e., at baseline and end of study. A referral mechanism will be followed for both intervention and control arm, which will ensure that the individuals with newly diagnosed diabetes will be referred to the nearest diabetes care facility.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Community mobilization will be done via male and female community groups using a PLA Cycle whereby groups themselves identify and priorities problems associated with diabetes and the risk of developing diabetes. Next this study will plan strategies to address the problems identified in the community, put these strategies into practice and, finally, evaluate the effectiveness of these strategies. Lay facilitators will convene the groups monthly over a period of 18 months, with one meeting per month.
  Interventions: Behavioral: Participatory, learning and Action (PLA) Based intervention
- Control Group (No Intervention): The Control Group will not receive the PLA (Participatory Learning and Action) intervention. However, they will still benefit from the study in several ways. Information about the trial and guidance on who to contact in case of hyperglycemia or intermediate hyperglycemia will be provided. The disease burden in the control area will be monitored, and findings will be included in national and international advocacy and dissemination efforts

INTERVENTIONS:
Behavioral: Participatory, learning and Action (PLA) Based intervention — An PLA based intervention would be carried out to prepare the Diabetes Mellitus type II patients. The intervention would be carried out for a tentative time of 2 to 3 hours to educate the type II diabetes mellitus. The study participants would be evaluated after completion of 18 months of the intervention. A structured, validated and literature-based assessment checklist will be devised to assess the effectiveness and feasibility of the intervention.
  Arms: Intervention Group

SUMMARY:
This project aims to adapt, implement, and evaluate PLA based intervention in urban Karachi, Pakistan for TIIDM prevention and control.

DETAILED DESCRIPTION:
The pivotal components of this approach include adapting, implementing, and evaluating the Participatory Learning and Action (PLA) based intervention for the prevention and control of Type II diabetes (TIIDM). TIIDM is considered the fastest-growing health emergency, affecting 537 million adults worldwide. Global projections for the year 2045 suggest that a 12.2% rise in TIIDM is anticipated with an additional 11.4% rise for intermediate hyperglycemia (IHG). Around 80% of people with TIIDM reside in low-and middle-income countries (LMICs), exhausting the already burdened healthcare system.

The intervention, adapted from the "Community groups or mobile phone messaging to prevent and control type 2 diabetes and intermediate hyperglycemia in Bangladesh (DMagic)" trial, has been tested and found effective in the rural context of Bangladesh. However, PLA-based intervention has not been previously tested in urban communities. Considering the distinct sociocultural environment of urban settings, a feasibility trial will be conducted in urban Karachi, Pakistan.

The feasibility trial will assess the intervention's adaptability and effectiveness in this new context. It is anticipated that the use of evidence-based approaches, best practices, and meaningful community participation through PLA will enhance the social and behavioral determinants of health and lead to improved health outcomes. This approach aims to control TIIDM and pave the way for managing other non-communicable diseases through similar focused interventions.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 20 years and above.
* Participants residing in the randomized clusters of Karachi, Pakistan
* Individuals willing to participate in the study and provide consent.
* Both individuals with normoglycemia, intermediate hyperglycemia, and diabetes are encouraged to participate.
* Participants who can attend the scheduled meetings and interventions as per the study protocol.

Exclusion Criteria:

* Individuals below the age of 20 years.
* Individuals unwilling to provide consent for participation.
* Participants with severe health conditions that may hinder their active involvement in the study.
* Individuals with non-compliance with research protocols

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 240 (Estimated)
Dates: Start 2024-06-24 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Type II Diabetes Mellitus | 18 months
  HbA1c biochemical test
Two-year cumulative incidence of Type II Diabetes Mellitus | 18 months
  HbA1c biochemical test

SECONDARY OUTCOMES:
Mean diastolic and systolic blood pressure | 18 months
  Digital blood pressure monitoring
Prevalence of hypertension | 18 months
  Digital BP monitoring
Abdominal obesity | 18 months
  Waist-to-hip circumference ratio
Mean body mass index | 18 months
  Height and weight will be taken
Health-related quality of life | 18 months
  World Health Organization Quality of Life (WHOQOL) BREF questionnaire
Frequency of depression | 18 months
  Patient Health Questionnaire (PHQ-9)
Mean body fat percentage | 18 months
  Using impedance analyzer
Prevalence of overweight and obesity | 18 months
  Height and weight will be taken
Frequency of anxiety | 18 months
  Generalized Anxiety Disorder (GAD-7) Scale

CONTACTS AND LOCATIONS:
Overall Officials: Abdul Basit, Director, Principal Investigator — Baqai Institute of Diabetes and Endocrinology
Locations (1):
- Baqai Institute of Diabetology and Endocrinology (BIDE), Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interested in the stated study area after its proper monitoring. Data or samples shared will be coded, with no PHI included. Prior permission of the investigators, participants and concerned departments will be obtained.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Data requests can be submitted starting 12 months after article publication
Access Criteria: Access can be requested by qualified researchers through proper approval of the investigators

REFERENCES:
- [Background] Imtiaz S, Khaleeq N, Sanauddin N, Afaq S, Jennings HM, Tahir A, Abdeali M, Khan Z, Khan F, Zafar R, Khan A, Shahab AR, Ali F, Elsey H, Hassan F, Khan A, Hofiani SMS, Alimi N, Azizi S, Alizoi N, Rahman K, Sheikh A, Basit A, Haq ZU. Community Health Participatory interventions in the prevention and control of non-communicable diseases including mental health in crisis-affected Low-and Middle-Income Countries - a scoping review. Glob Health Action. 2026 Dec;19(1):2599011. doi: 10.1080/16549716.2025.2599011. Epub 2026 Jan 2. PMID 41480977
- [Derived] Imtiaz S, Zafar R, Tahir A, Abdeali M, Ahmed F, Mansoor A, Khan A, Fawwad A, Basit A, Walker S, Afaq S, Rehman K, Khan Z, Kanaan M, Jennings HM, Shahab AR, Siddiqi K, Haq ZU. Engagement of coMmunity through Participatory learning and action for cOntrol and preVEntion of Type 2 Diabetes and its Risk factors (EMPOWER-D): protocol for a feasibility cluster randomised controlled trial in urban Pakistan. Pilot Feasibility Stud. 2026 Feb 3. doi: 10.1186/s40814-025-01762-x. Online ahead of print. PMID 41630102
- See also: OSF registration link — https://doi.org/10.17605/OSF.IO/EU95B